CLINICAL TRIAL: NCT06285695
Title: Clareon Toric Single Arm Study (T2-T9)
Brief Title: Clareon Toric Study (T2-T9)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILS241-I001
Record Dates: First submitted 2024-02-23; First posted 2024-02-29 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Aphakia; Corneal Astigmatism
MeSH Terms: conditions — Aphakia; Astigmatism | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Clareon Toric IOL (Experimental): Clareon Toric IOL implanted in one or both eyes during cataract surgery
  Interventions: Device: Clareon Toric IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: Clareon Toric IOL — Aspheric hydrophobic acrylic IOL placed in the capsular bag in the posterior chamber of the eye during cataract surgery for the visual correction of aphakia and preexisting corneal astigmatism
  Other Names: Models CNW0T2, CNW0T3, CNW0T4, CNW0T5, CNW0T6, CNW0T7, CNW0T8, CNW0T9, CNA0T2, CNA0T3, CNA0T4, CNA0T5, CNA0T6, CNA0T7, CNA0T8, CNA0T9
Procedure: Cataract surgery — Cataract extraction by phacoemulsification, followed by implantation with a Clareon Toric IOL

SUMMARY:
The purpose of this post-market study is to describe the long-term safety and performance of Clareon Toric Intraocular Lenses (IOLs).

DETAILED DESCRIPTION:
Subjects will attend up to 12 scheduled visits (one preoperative visit, up to two surgical visits, and up to 9 postoperative visits) over the course of the study (3 years follow-up). The overall study duration is expected to be approximately 4 years. This study will be conducted in Canada.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign the informed consent form.
* Willing and able to attend all scheduled study visits as required per protocol.
* Cataract in one or both eyes with planned extraction by conventional phacoemulsification.
* Astigmatism in the operative eye(s).
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Women of childbearing potential, currently pregnant, intend to become pregnant during the study, or nursing.
* History of retinal detachment, age-related macular degeneration, glaucoma, diabetic retinopathy, or any pathologic changes associated with the optic nerve.
* Clinically significant corneal disease that may, according to the Investigator's medical opinion, adversely affect visual outcomes.
* Clinically significant dry eye that would affect study measurements based on the Investigator's expert medical opinion.
* History of prior intraocular or corneal surgery.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Mean monocular best corrected distance visual acuity (BCDVA) | Month 6, Year 1, Year 3 (post implantation)
  Visual acuity will be assessed for each eye individually using letter charts and recorded in logarithm minimum angle of resolution (logMAR).

SECONDARY OUTCOMES:
Mean monocular absolute residual refractive cylinder | Month 3, Month 6, Year 1, Year 3 (post implantation)
  The amount of residual astigmatism will be assessed for each eye individually using letter charts and recorded in diopters.
Mean absolute IOL rotation from previous visit | Month 1 to Month 3, Month 3 to Month 6, Month 6 to Year 1, Year 1 to Year 3 (post implantation)
  The difference in IOL axis of orientation from the previous visit will be assessed by a reading center and recorded in degrees.
Mean absolute IOL rotation from end of surgery supine baseline to each subsequent visit | Baseline, Day 1, Week 1, Month 1, Month 3, Month 6, Year 1, Year 3 (post implantation)
  The difference in IOL axis of orientation from baseline (end of surgery, patient laying flat) will be assessed by a reading center and recorded in degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management Operations, Surgical, Study Director — Alcon Research, LLC
Locations (6):
- Canada (6):
  - Gimbel Eye Centre, Calgary, Alberta
  - Uptown Eye Specialists, Concord, Ontario
  - Prism Eye Institute, Oakville, Ontario
  - Laurentians Eye Institute, Boisbriand, Quebec
  - Bellevue, Montreal, Quebec
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No